CLINICAL TRIAL: NCT03819140
Title: Continuous Versus Cyclical OCP Use in PCOS: A Pilot Study
Brief Title: Continuous Versus Cyclical OCP Use in PCOS
Acronym: CCOUP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-24705
Record Dates: First submitted 2018-11-29; First posted 2019-01-28 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Hyperandrogenism; Oral Contraceptive Pills
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continuous OCP Therapy (Active Comparator): Participants randomly assigned to this arm will receive 8 packs of a 21 day oral contraceptive pills (OCP) called Yasmin (3 mg Drospirenone/0.03 mg Ethinyl estradiol) which comes in a formulation of 21 days of active hormone and 7 days of sugar pills. In this arm, participants will only be expected to take active hormone pills (colored pills) for the 6 months straight without stopping or taking the sugar pills in each pack.
  Interventions: Drug: Yasmin
- Cyclical OCP Therapy (Active Comparator): Participants randomly assigned to this arm will receive 6 packs of a 21 day oral contraceptive pill (OCP) called Yasmin (3 mg Drospirenone/0.03 mg Ethinyl estradiol) which has 21 days of active hormone and 7 days of sugar pills. Participants will take one pill daily for 6 months and be expected to take the sugar pills at the end of each monthly pack prior to starting a new pack.
  Interventions: Drug: Yasmin

INTERVENTIONS:
Drug: Yasmin — Participants in each treatment arm will receive the medication Yasmin. However only the Cyclical OCP Therapy arm will take the sugar pills designated each month in the pill packs and the Continuous OCP Therapy arm will not.

SUMMARY:
The mainstay treatment for females with Polycystic Ovary Syndrome (PCOS) has long been a combination of an oral contraceptive pill or OCP (containing both estrogen and progestin) along with an anti-androgen medication (such as Spironolactone) to not only prevent chronic anovulation but also suppress elevated testosterone levels and its clinical effects on the body. While there are multiple OCPs available on the market today and several studies that look at different progestins and their anti-androgenicity, not much is known about whether the length of active pills in OCP therapy (3 weeks versus 6 months) has any further benefit in continued suppression of testosterone and subsequently improvement in clinical findings of hyperandrogenism in the PCOS population. In this pilot randomized open label clinical trial, females between the ages of 16 and 35 years diagnosed with PCOS based on the Rotterdam Criteria, and not currently on medical therapy with an OCP will be enrolled in the study and randomized to either a continuous 6 month OCP or cyclical 21 day active OCP therapy. Our aim is to conduct a pilot randomized clinical trial to determine the effect of 6 months of active monophasic OCPs on testosterone levels and cutaneous findings of hyperandrogenism (hirsutism and acne) as compared to a traditional 21 day active/7 day placebo OCP in women with PCOS. These findings will be compared over a 6 month period.

DETAILED DESCRIPTION:
Those who meet criteria to take part in the study (women between the ages of 16-35 years, diagnosed with PCOS and have findings of hyperandrogenism either by serum testosterone levels above the normal reference range or by their modified Ferriman Gallwey score of >8, and are recommended to start an oral contraceptive pill for therapy) and give consent, will be randomized into either of two oral contraceptive (OCP) treatment groups:

1. Ethinyl estradiol 30 mcg-Drospirenone 3 mg (Yasmin): 168 days of active hormone pills (no placebo pills) for 6 months.
2. Ethinyl estradiol 30 mcg-Drospirenone 3mg (Yasmin): 21 days of active + 7 days of placebo pills for 6 months

Participants will be given the OCP Yasmin with instructions to take the medication at the same time each day for the length of the study (6 months). On the 4th, 12th and 24th week of therapy (roughly the 1st, 3rd and 6th month), blood work will be drawn and is detailed below.

At 1 month into therapy, (near the end of the 4th week on an OCP) both treatment groups will be expected to get blood work (total and free testosterone, SHBG, estradiol, LH, and FSH levels will be checked). At the time of the blood draw, subjects in the cyclical group should be on placebo/sugar pills and those in the continuous group on active hormone pills.

At 3 months into therapy, participants will come back to the PCOS clinic for routine care follow up and be seen by a Reproductive Endocrinology and Fertility specialist. This visit is considered "standard of care" and not specific to the study. However, during this visit a study investigator will also touch base briefly with the participants to see how they are doing. An online survey (through REDCap) will also be sent to participants that addresses if they have missed any doses of their medication and assess their acne quality of life. In addition, participants will once again get blood work (including total and free testosterone, SHBG, estradiol, LH, FSH, fasting lipid panel, fasting serum glucose, insulin, and HbA1c). As before, the cyclical group should be on placebo/sugar pills at the time of blood draw and the continuous group on active hormone pills.

At 6 months into therapy, participants will come in for a study visit (this is not considered routine care) in which they will have their vitals taken, a physical exam that includes a re-evaluation of their mFG score, and an in-clinic pelvic ultrasound to assess ovarian volume and follicle counts. They will also be emailed a post-study survey through REDCap, that includes a quality of life questionnaire for both acne and hirsutism, and includes questions regarding satisfaction with current therapy and any missed doses of their medication. Lastly, participants will again be expected to get blood work (total and free testosterone, SHBG, estradiol, LH, FSH).

ELIGIBILITY:
Inclusion Criteria: To be included in this study, participants must be:

1. Female, within 15-40 years of age
2. Diagnosed with Polycystic Ovary Syndrome based on the 2003 Rotterdam Criteria (must meet 2 out of 3 criteria):

   1. evidence of either biochemical or clinical hyperandrogenism (elevated free and or total testosterone level above the normal reference range for assay, and/or an modified Ferriman-Gallwey hirsutism score >8)
   2. Oligo- or anovulation
   3. Polycystic ovary morphology on ultrasound
3. Adolescents should be at least 2 years out from menarche (first menstrual period).
4. Participants must not be on an oral contraceptive pill (OCP) at the start of the study and or Spironolactone therapy (an anti-androgen medication), but recommended by their physician to start OCP therapy.

Exclusion Criteria:

1. Females with Polycystic Ovary Syndrome (PCOS) who do not have either biochemical (elevated total or free testosterone levels) or clinical (modified Ferriman-Gallwey hirsutism score <8) findings of hyperandrogenism will not be included in the study as this is one of the primary outcome measures.
2. Females with PCOS who are already on and currently using a form of contraceptive (oral, vaginal ring, or patch)
3. Females that are concurrently using or plan to use an anti-androgenic medication such as Spironolactone in the next 6 months.
4. Females currently or are planning to obtain permanent hair removal (ex. laser hair removal, electrolysis) in the concurrent 6 months of starting oral contraceptive (OCP) therapy will also be excluded from the study
5. Women who are pregnant or have contraindications for starting an OCP, including active smokers, history of clotting disorders, history of deep vein thrombosis or blood clots, neoplasia, vascular disease, migraines, hypertension, or have renal/hepatic disease will be excluded from the study as OCP therapy would not be indicated or approved in this population.
6. Females with elevated potassium levels above the normal reference range for age.

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legro RS, Pauli JG, Kunselman AR, Meadows JW, Kesner JS, Zaino RJ, Demers LM, Gnatuk CL, Dodson WC. Effects of continuous versus cyclical oral contraception: a randomized controlled trial. J Clin Endocrinol Metab. 2008 Feb;93(2):420-9. doi: 10.1210/jc.2007-2287. Epub 2007 Dec 4. PMID 18056769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between April 2019 and January 2022 at the UCSF Center for Reproductive Health's PCOS multidisciplinary clinic.
Period: Overall Study
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
Started | 26 | 25
1 Month on Yasmin | 21 | 21
3 Months on Yasmin | 19 | 19
6 Months on Yasmin | 19 | 16
Completed | 19 | 16
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Unable to attend visit(s) due to contracting COVID | 2 | 1
Not completed — Unable to attend visit(s) due to UCSF pandemic policies restricting non-essential visits | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 16 | 10 | 26
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51
Serum Total Testosterone [Mean (Standard Deviation); unit: ng/dl] | 32.4 (15.3) | 29.5 (18.5) | 30.97 (16.94)
Modified Ferriman-Gallwey (mFG) score [Mean (Standard Deviation); unit: units on a scale] | 13 (5) | 14 (7) | 13.49 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Biochemical Hyperandrogenism From Baseline to 1 Month Post Yasmin Initiation
Description: Positive or negative change in blood serum Total Testosterone value (units: ng/dl) from baseline to 1 month post Yasmin initiation.
Time Frame: measured at baseline and 1 month into therapy
Population: Analysis exclusions: 1 non-compliant initially with taking continuous dose, 1 unable to promptly obtain yasmin from pharmacy, 1 unresponsive to appointment scheduling reminders, 6 insufficient specimen volume to run assay and unable to calculate change value.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
Number analyzed (Participants) | 21 | 21
ng/dl | -15.38 (13.15) | -8.54 (17.66)

2. Primary Outcome: Change in Biochemical Hyperandrogenism From Baseline to 3 Month Post Yasmin Initiation
Description: Positive or negative change in blood serum Total Testosterone value (units: ng/dl) from baseline to 3 month post Yasmin initiation.
Time Frame: measured at baseline and 3 month into therapy
Population: Analysis exclusions: 3 unable to attend appointment due to COVID, 3 participants elected to drop out of study as desired to switch to another brand of OCP, 3 participants were unresponsive to communications to schedule appointment. 4 contracted COVID or unable to attend visit due to UCSF restriction on non-essential visits during COVID lockdown
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
Number analyzed (Participants) | 19 | 19
ng/dl | -17.05 (17.13) | -4.58 (16.46)

3. Primary Outcome: Change in Biochemical Hyperandrogenism From Baseline to 6 Month Post Yasmin Initiation
Description: Positive or negative change in blood serum Total Testosterone value (units: ng/dl) from baseline to 6 month post Yasmin initiation.
Time Frame: measured at baseline and 6 month into therapy
Population: Analysis exclusions (16): 3 voluntarily dropped out of study for personal reasons, 3 unresponsive to appointment scheduling reminders,1 broke fast and unable to draw, 1 specimen hemolyzed and unable to run assay, 4 contracted COVID or unable to attend visit due to UCSF restriction on non-essential visits during COVID lockdown,4 insufficient specimen volume to run 6 month assay and unable to calculate change value.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
Number analyzed (Participants) | 19 | 16
ng/dl | -13.53 (19.25) | -9.36 (13.29)

4. Secondary Outcome: Change in Clinical Findings of Hyperandrogenism - Hirsutism
Description: Participants will be examined by a physician and scored using the modified Ferriman-Gallwey Hirsutism score (mFG). This scoring system is considered the standard scoring system that defines hirsutism (excess male pattern hair growth on the body) quantitatively. There are 9 body areas measured on a scare of 0-4, with higher values indicative of significant hair growth. All subscales are combined for a total score, with a minimum score of 0 and max of 36. A total score of >/=8 is considered diagnostic for hirsutism. The difference in score values from baseline to 6 months was then calculated.
Time Frame: Baseline and at 6 months into therapy
Population: Analysis exclusions: 8 of the 35 participants who attended the 6 month visit declined the physical exam necessary for physician mFG scoring and thus changes in mFG scores from baseline to 6 months could not be calculated for these participants.
Measure: Mean (Standard Deviation); unit: numerical change in score on a scale
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
Number analyzed (Participants) | 14 | 13
numerical change in score on a scale | -3.14 (2.85) | -1.62 (3.36)

5. Secondary Outcome: Metabolic Changes With OCP Therapy
Description: Diabetes risk will be assessed and compared in both treatment arms by measuring HOMA-IR (calculated as [glucose*insulin]/405) at both baseline and 3 months visits and calculating the change in HOMA-IR value. Higher HOMA-IR values indicate more severe insulin resistance, with the ranges being as follows: HOMA <2: Normal, HOMA 2-4: Mild Insulin Resistance, and HOMA >4: Moderate-Severe Insulin Resistance.
Time Frame: Baseline and at 3 months into therapy
Measure: Mean (Standard Deviation); unit: HOMA-IR value
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
Number analyzed (Participants) | 19 | 19
HOMA-IR value | 0.007 (0.130) | 0.071 (0.269)

ADVERSE EVENTS:
Time Frame: 6 months while on Yasmin
Arm/Group | Continuous OCP Therapy | Cyclical OCP Therapy
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous OCP Therapy (N=26) | Cyclical OCP Therapy (N=25)
Undisclosed Exclusion Criteria - Symptoms and History of Migraines with Aura (Nervous system disorders) | 0 (0) | 1 (1) — More serious than expected, possibly related to study. PI removed the participant from the study by having her stop the OCP due to the severe migraines with aura that she was having on 2/2/2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03819140/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03819140/ICF_001.pdf